CLINICAL TRIAL: NCT04834050
Title: Can 4 Weeks of Exercise Program Change Quadriceps Architecture in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ovgu Bickici (Other Government)
Responsible Party: Sponsor-Investigator, Ovgu Bickici, OB, Hatay Dortyol State Hospital
Organization: Hatay Dortyol State Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26022019
Record Dates: First submitted 2021-03-31; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Arthritis, Rheumatoid; Knee Osteoarthritis; Quadriceps Muscle Atrophy; Ultrasonography; Exercise
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rheumatoid arthritis patients (Experimental)
  Interventions: Procedure: Quadriceps femoris isometric home-based exercise
- Knee Osteoarthritis patients (Experimental)
  Interventions: Procedure: Quadriceps femoris isometric home-based exercise
- Healthy patients (Experimental)
  Interventions: Procedure: Quadriceps femoris isometric home-based exercise

INTERVENTIONS:
Procedure: Quadriceps femoris isometric home-based exercise — All 3 groups of participants were given 4-week (5 days/week) quadriceps-hamstring isometric home-based exercise training for their both knees. Exercises were performed (with maximal effort for 10 seconds) at a rate of 20 repetitions per day. Training was performed at outpatient clinic for 30 minutes.

SUMMARY:
Quadriceps femoris (QF) atrophy is seen in rheumatoid arthritis and knee osteoarthritis (OA) patients. Exercise therapy is mile stone in knee OA patients also it can help thicken QF muscle of RA patients. We primarily aimed to demonstrate the influence of 4 weeks of knee isometric home-based training on QF muscle parts thickness and pennation angle measurements of RA patients with ultrasonography (USG). This study included 12 patients with RA, 12 patients with knee OA as positive control group and 13 volunteers as healthy control group. All participants were given 4 weeks of quadriceps-hamstring isometric home-based training. At baseline and at the end of the program, WOMAC and Lequesne algofunctional index scores of knee OA patients and DAS28-CRP scores of RA patients were recorded. Dominant knee thickness and pennation angle measurements of QF muscle parts were evaluated by ultrasonography.

ELIGIBILITY:
The inclusion criteria for all participants were being between 18-65 yy.

The inclusion criteria for RA patients were: confirmed diagnosis of RA according to 2010 ACR/EULAR classification criteria and lack of any other inflammatory articular diseases.

The inclusion criteria for knee OA patients were: diagnosis according to ACR classification criteria of knee OA with grade 2-3 according to the Kellgren-Lawrence grading system and lack of any other inflammatory articular diseases.

Volunteers who did not have any knee pain, no clinical degenerative or inflammatory signs were included in the healthy control group.

-

Exclusion criteria for all participants were: being out of age range, history of knee joint trauma, surgery or knee joint injection in the previous 6 months, presence of any other disease that can affect thigh muscles (radiculopathy, myopathy, hip problems). Patients with secondary knee OA were not included.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Change of quadriceps femoris parts thickness measures | At baseline and after 4 weeks of intervention
  Dominant knee vastus lateralis, medialis, intermedius and rectus femoris thicknesses of 3 groups were calculated at baseline and at the end of intervention.
Change of quadriceps femoris parts pennation angles | At baseline and after 4 weeks of intervention
  Pennation angles of vastus lateralis, medialis and intermedius were calculated at baseline and at the end of exercise program.

SECONDARY OUTCOMES:
Change of The Western Ontario and McMaster Universities Arthritis Index (WOMAC) score of knee OA | At baseline and after 4 weeks of intervention
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) scores of knee OA patients were calculated at baseline and at the end of exercise program. The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is divided into 3 subscales: Pain, stiffness, physical function. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of scores of 3 subscales were multipled with 100 and divided by 96 and resulted in WOMAC score of the patients.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Change of Disease activity score 28-C reactive protein (DAS28-CRP) | At baseline and after 4 weeks of intervention
  Disease activity score 28-C reactive protein (DAS28-CRP) scores of RA patients were calculated at baseline and at the end of program. A score lower than 2.6 means remission, score between 2.6 and 3.2 means low disease activity, score between 3.2 and 5.1 means moderate disease activity and score higher than 5.1 means high disease activity.
Change of Lequesne scores of knee OA patients | At baseline and after 4 weeks of intervention
  Lequesne algofunctional index scores of knee OA patients were calculated at baseline and at the end of the intervention. The Lequesne OA index is scored as the sum of questions ranging from 0 to 24, higher scores meaning worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No